CLINICAL TRIAL: NCT01476657
Title: A Phase 1 Study of Duvelisib in Patients With Advanced Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The scope of the program has been reduced to focus resources on studies which can potentially enable the registration of duvelisib.
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-145-02
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hematologic Malignancies
Keywords: Phase 1
MeSH Terms: conditions — Hematologic Neoplasms | interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-145 (Experimental): IPI-145 is administered orally as a capsule formulation. The IPI-145 drug product is supplied as 1 mg, 5 mg, 25 mg, and 100 mg formulated capsules. IPI-145 will be administered orally daily during each 28-day cycle. Patients will be evaluated for DLTs in the dose escalation portion of the study during Cycle 1 (28 days), after which treatment may continue for additional cycles.
  Interventions: Drug: IPI-145 (duvelisib)

INTERVENTIONS:
Drug: IPI-145 (duvelisib) — Oral Twice A Day (BID) Dosing

SUMMARY:
The purpose of this study is to determine the safety, maximum tolerated dose and pharmacokinetics of IPI-145 in patients with advanced hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age;
* Progressed during, refractory to, intolerant of, or ineligible for established therapy, or has a disease with no established therapy with the exception of expansion cohort of treatment naïve CLL patients;
* An Eastern Cooperative Oncology Group (ECOG) score of 0 to 2.

Exclusion Criteria:

* Any previous treatment with a PI3K inhibitor (Escalation Phase only) or within 4 weeks of the start of IPI-145 administration (Expansion Phase);
* Patients with overt leptomeningeal leukemia or CNS lymphoma;
* Inadequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN); direct bilirubin >1.5 x ULN;
* Inadequate renal function defined by serum creatinine > 1.5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-10; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | At least 28 days (1 Cycle)
  To determine the incidence of adverse events and abnormal laboratory test results, including dose-limiting toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (4):
- United States (4):
  - New York, New York
  - Columbus, Ohio
  - Nashville, Tennessee
  - Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Horwitz SM, Koch R, Porcu P, Oki Y, Moskowitz A, Perez M, Myskowski P, Officer A, Jaffe JD, Morrow SN, Allen K, Douglas M, Stern H, Sweeney J, Kelly P, Kelly V, Aster JC, Weaver D, Foss FM, Weinstock DM. Activity of the PI3K-delta,gamma inhibitor duvelisib in a phase 1 trial and preclinical models of T-cell lymphoma. Blood. 2018 Feb 22;131(8):888-898. doi: 10.1182/blood-2017-08-802470. Epub 2017 Dec 12. PMID 29233821
- [Derived] Flinn IW, O'Brien S, Kahl B, Patel M, Oki Y, Foss FF, Porcu P, Jones J, Burger JA, Jain N, Kelly VM, Allen K, Douglas M, Sweeney J, Kelly P, Horwitz S. Duvelisib, a novel oral dual inhibitor of PI3K-delta,gamma, is clinically active in advanced hematologic malignancies. Blood. 2018 Feb 22;131(8):877-887. doi: 10.1182/blood-2017-05-786566. Epub 2017 Nov 30. PMID 29191916
- [Derived] Patel VM, Balakrishnan K, Douglas M, Tibbitts T, Xu EY, Kutok JL, Ayers M, Sarkar A, Guerrieri R, Wierda WG, O'Brien S, Jain N, Stern HM, Gandhi V. Duvelisib treatment is associated with altered expression of apoptotic regulators that helps in sensitization of chronic lymphocytic leukemia cells to venetoclax (ABT-199). Leukemia. 2017 Sep;31(9):1872-1881. doi: 10.1038/leu.2016.382. Epub 2016 Dec 26. PMID 28017967